CLINICAL TRIAL: NCT00630097
Title: A Dose Ranging Study of Modafinil for Methamphetamine Dependence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Gantt Galloway, California Pacific Medical Center Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27.140
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Substance Dependence; Amphetamine Dependence
Keywords: methamphetamine addiction, meth dependence
MeSH Terms: conditions — Substance-Related Disorders; Amphetamine-Related Disorders | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: modafinil — Modafinil, 100mg, 400mg, or 600 mg tablets QD for 4 weeks.

SUMMARY:
Patients treated for methamphetamine dependence have high rates of relapse, and no pharmacotherapy has yet been demonstrated to be efficacious. Modafinil (d, l-2-[(diphenylmethyl)sulfinyl]acetamide) is a novel wake- and vigilance-promoting agent that is chemically and pharmacologically dissimilar to CNS stimulants. It is well tolerated and has low abuse liability compared to CNS stimulants. Modafinil is FDA approved for a variety of sleep disorders, may relieve methamphetamine withdrawal symptoms, improves cognitive function, has been shown to reduce cocaine use in dependent users, and is safe when coadministered with intravenous methamphetamine. We will conduct a randomized dose ranging clinical trial of modafinil to establish its safety and efficacy as a pharmacotherapy for methamphetamine dependence.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50 years
2. Patient is agreeable to conditions of study and signs consent form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Methamphetamine-negative urine samples will be analyzed using a generalized estimating equation model | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Gantt Galloway, PharmD, Principal Investigator — California Pacific Medical Center
Locations (1):
- CPMC, San Francisco, California, United States